CLINICAL TRIAL: NCT02327572
Title: Age-related Changes in the Immune System and Their Impact on Elderly Breast Cancer
Acronym: IMAGE
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjunct head of clinic, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56278 UGasthuisberg; S56278 (Other Grant/Funding Number: stichting tegen kanker); NCT02176447 (obsolete NCT alias)
Record Dates: First submitted 2014-12-08; First posted 2014-12-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (two 10-mL EDTA tubes) will be collected from each patient immediately prior to surgery for assessing ageing/immunosenescence biomarkers
Oversight: Data Monitoring Committee: No

SUMMARY:
This research project aims to study this intriguing relationship between ageing and breast cancer biology, and more specifically the changes that occur within the tumor microenvironment with increasing age. Furthermore, it will focus on the link between these microenvironmental changes and organismal ageing (as measured by chronological age, geriatric evaluation of elderly patients, and circulating biomarkers of ageing), since it seems logical that age-related changes in the stromal part of a tumor (fibroblasts, immune cells, endothelial cells, fatty cells, …i.e. host cells) are due to the ageing process of the entire body. Most particularly, the amount and type of infiltrating immune cells might reflect the degree of immunosenescence of the host. More and more research points out the crucial role of the immune system in tumorigenesis and progression, and, at the same time, the immune system is one of the most affected components in the process of ageing. .

DETAILED DESCRIPTION:
Despite the high relevance of ageing/immunosenescence and frailty in oncogeriatric practice, immuno-senescence markers have so far not been considered in concert with clinical tumor characteristics and the profile of tumor infiltrating leukocytes. In the proposed project, the investigators will examine immunosenescence markers in blood and characterize the leukocyte infiltrate in the tumor microenvironment in the setting of elderly breast cancer.

The main goal of this project is thus to investigate the relation and interaction between the following 3 aspects:

(i) immune status of the host: chronological age and immunosenescence in peripheral blood; (ii) tumor microenvironment: local immune response (evaluated via assessment of the amount and nature of tumor infiltrating leukocytes [TIL]); (iii) clinical tumor characteristics: tumor size, grade, receptor status, lymph node involvement.

To realize this project, the investigators will set up a prospective clinical study comprising three distinct age categories of breast cancer patients and integrating a variety of immunosenescence markers. Different specific manifestations of immune system ageing will be studied : age-related pro-inflammatory status (inflammageing), increased expression of the senescence marker p16INK4a in T lymphocytes, shifts in subset composition of the PBMC pool, age-associated changes in expression of immune-related genes in PBMC and altered abundance of specific ageing-related plasma microRNAs.

At the tumor microenvironmental level, the leukocyte infiltrate will be studied in detail. The profile of tumor-infiltrating immune cells will be compared between the distinct age groups and will be correlated to systemic markers of ageing/immunosenescence (in blood) and tumor biology, most particularly lymph node involvement.

Concrete research questions:

* How are the different immunosenescence markers (i.e. subset profile of PBMC, pro-inflammatory markers in plasma, lymphocyte senescence as evidenced by p16INK4a expession in T lymphocytes, expression of immune-related genes in PBMC and abundance of ageing-related circulating microRNAs) correlated with each other and with the patient's calendar age?
* Does the local immune response in the tumor (amount and nature of TIL) correlate with the different immunosenescence markers?
* Is there a relationship between tumor biology, most particularly lymph node involvement, and the local immune response in the tumor ?

With this study, the investigators intend to improve our fundamental understanding of age-related changes in general immune status and tumor-specific immune responses and their impact on tumor progression. This may add to recent advances in newly emerging therapeutic strategies, such as immune-related approaches. Due to recent advances in biology and genomics, it has become possible to personalize an individual's cancer treatment based on molecular tumor characteristics. In the elderly, however, host factors also become increasingly important and may influence both tumor behavior/progression and therapy tolerance/response. Therefore, a better understanding of the biological mechanisms underlying ageing/immunosenescence, its association with cancer and the potential prognostic/predictive information that the patient's ageing/immunosenescence profile can provide is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* o Patients newly diagnosed with breast cancer who will undergo surgery and gave written informed consent

  * Group 1 : 30 patients aged 70+ Group 2 : 15 patients aged 55-65 (post-menopausal) Group 3 : 15 patients aged 35-45 (pre-menopausal)
  * Tumor selection : grade II/III invasive tumor, any histological type, ER-positive, HER2-negative
  * Tumor size ≥1.5 cm (clinical assessment: mammoechography and/or clinical examination)

Exclusion Criteria:

-

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients newly diagnosed with breast cancer who will undergo surgery and gave written informed consent
  * Group 1 : 30 patients aged 70+ Group 2 : 15 patients aged 55-65 (post-menopausal) Group 3 : 15 patients aged 35-45 (pre-menopausal)
  * Tumor selection : grade II/III invasive tumor, any histological type, ER-positive, HER2-negative
  * Tumor size ≥1.5 cm (clinical assessment: mammoechography and/or clinical examination)
  * Routine geriatric assessment performed prior to surgery in group 1.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
- Are there differences in tumor stroma, both with regard to immune infiltration and cellular senescence, between young and old patients, and between old fit and old frail patients? | at diagnosis

SECONDARY OUTCOMES:
- Does the local immune response in the tumor (amount and type of infiltrating cells) correlate with subset profile of circulating immune cells (PBMC) and immunosenescence markers in the plasma, and with clinical ageing? | at diagnosis
- Is there a relation between senescence markers expressed in tumor stroma (SAβ-galactosidase, heterochromatinisation, SASP) and ageing markers measured in the blood? | at diagnosis
- Do immune infiltration of the tumor, stromal senescence in the tumor and plasma ageing/immunosenescence profile correlate with relapse and survival (long term outcome)? | at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: hans wildiers, Study Chair — department of general medical oncology
Locations (1):
- University Hospitals Leuven, Leuven, Belgium